CLINICAL TRIAL: NCT00512694
Title: Duke Lupus Registry
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00008875; 8652-07-6R1 (Other: Duke legacy protocol number)
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus; Cutaneous Lupus
Keywords: Lupus; Systemic Lupus Erythematosus; Cutaneous Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for future research.
Oversight: Data Monitoring Committee: No

SUMMARY:
Lupus is a systemic autoimmune disease that can present with many varied symptoms, including joint pain, fevers, kidney disease, and rashes. Lupus can affect anyone, but it is most common in younger women.

The Duke Lupus Registry will collect information and blood samples from patients with lupus (systemic lupus erythematosus or cutaneous lupus) seen in the Duke Rheumatology clinics. The goal of this Registry is to understand how lupus changes over time so that we can improve the treatment of patients with lupus.

DETAILED DESCRIPTION:
The Duke Lupus Registry is a prospective cohort comprised of patients with lupus seen in the Duke Rheumatology clinic.

The Duke Lupus Registry has two main purposes:

1. Improved patient care. By following disease activity scores and medication usage, we expect to improve our care of the patients seen in clinic.
2. Future research on lupus outcomes. This may encompass a broad array of areas, including but not limited to cardiovascular health, pregnancy and fertility, infections, medication use, quality of life, and depression.

At each office visit, patients will complete a questionnaire, physicians will measure lupus activity, and patients may be asked to provide a small blood sample. Patients will not be required to make extra visits to Duke in order to participate -- all paperwork and blood draws will occur during a regularly scheduled office visit with the physician.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Systemic Lupus Erythematosus or Cutaneous Lupus
* Patient of a rheumatologist at Duke University Medical Center

Exclusion Criteria:

* Inability to travel to Duke for follow-up visits
* Inability to speak English
* Not able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients with lupus.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-07; Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Megan E. B. Clowse, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- See also: The Duke Lupus Clinic website — http://www.dukehealth.org/locations/duke_lupus_clinic